CLINICAL TRIAL: NCT01255748
Title: Evaluation Tracking Project: A Prospective Chart Review of Patients Treated With Radiation Therapy
Brief Title: Registry Study for Radiation Therapy Outcomes
Status: Recruiting | Type: Observational
Sponsor: Proton Collaborative Group (Network)
Responsible Party: Sponsor
Other Study IDs: REG001-09
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms
Keywords: cancer, proton, radiation
MeSH Terms: conditions — Neoplasms | interventions — Proton Therapy; Spermine Synthase; Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment with Radiation Therapy: Includes 16 different arms to capture patient data by disease site
  Interventions: Radiation: Proton Therapy, Photon Therapy, SRS, Brachytherapy

INTERVENTIONS:
Radiation: Proton Therapy, Photon Therapy, SRS, Brachytherapy — Outcomes Tracking

SUMMARY:
The purpose of this research study is to collect and analyze information from patients being treated with various forms of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Planned treatment with radiation therapy
* Ability to understand and sign IRB approved consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Radiation Oncology patients
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2009-06; Primary Completion 2039-06 (Estimated)

PRIMARY OUTCOMES:
Define outcomes for patients treated at participating institutions | PRN

SECONDARY OUTCOMES:
Determine strategies necessary to improve patients outcome and decrease toxicities related to treatments and procedures | Annually PRN
Improve patient care by an adequate understanding of the results and patient population at participating institutions | Reviewed Annually PRN

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Vargas, MD, Study Chair — Proton Collaborative Group
Locations (29):
- United States (29):
  - Mayo Clinic, Scottsdale, Arizona
  - Proton Center of Arkansas, Little Rock, Arkansas
  - California Protons Cancer Therapy Center, San Diego, California
  - South Florida Proton Therapy Institute, Delray Beach, Florida
  - Ackerman Cancer Center, Jacksonville, Florida
  - Dwoskin Proton Therapy Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - OSF HealthCare Cancer Institute, Peoria, Illinois
  - Northwestern Medicine Chicago Proton Center, Warrenville, Illinois
  - University of Kansas Proton Therapy Center, Kansas City, Kansas
  - Kansas City Proton Institute, Overland Park, Kansas
  - Willis-Knighton Cancer and Proton Therapy Center, Shreveport, Louisiana
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - McLaren Proton Therapy Center, Flint, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Mercy David C. Pratt Cancer Center, St Louis, Missouri
  - ProCure Proton Therapy Center, Somerset, New Jersey
  - New York Proton Center, New York, New York
  - Atrium Health Levine Cancer Proton & Advanced Radiation Center, Charlotte, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oklahoma Proton Center, Oklahoma City, Oklahoma
  - Tennessee Oncology Proton Center, Franklin, Tennessee
  - Thompson Proton Center, Knoxville, Tennessee
  - Texas Center for Proton Therapy, Irving, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Hampton University Proton Therapy Institute, Hampton, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Lee HJ Jr, Macomber MW, Spraker MB, Bowen SR, Hippe DS, Fung A, Russell KJ, Laramore GE, Rengan R, Liao J, Apisarnthanarax S, Zeng J. Early toxicity and patient reported quality-of-life in patients receiving proton therapy for localized prostate cancer: a single institutional review of prospectively recorded outcomes. Radiat Oncol. 2018 Sep 17;13(1):179. doi: 10.1186/s13014-018-1127-6. PMID 30223877
- See also: Sponsor's website — http://www.pcgresearch.org